CLINICAL TRIAL: NCT00638417
Title: Treatment and Rehabilitation of Patients With Hip Arthroplasty to Regain Walk and Work Efficiency and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: OrtoMedic A/S, Oslo (Unknown); Scandinavian Customized Prosthesis (SCP) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2005.1527a
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maximal strength training (Experimental): maximal dynamic strength training
  Interventions: Behavioral: Maximal strength training; Behavioral: conventional rehabilitation
- conventional rehabilitation (Other): rehabilitation as usual
  Interventions: Behavioral: conventional rehabilitation

INTERVENTIONS:
Behavioral: Maximal strength training — maximal dynamic strength training from 1 week after the operation, 5 training bouts a week for 4 weeks. The regimen consisted of 2 exercises, leg press and hip abduction, that included 4 series of 5RM involving the operated leg only. 5RM corresponds to approximately 85% of 1RM. When the patients managed to perform 6RM, the load was increased by 5kg. The series were separated by resting periods of 2 minutes.
  Arms: maximal strength training
Behavioral: conventional rehabilitation — conventional rehabilitation program: inpatient treatment in a rehabilitation center. Individual sling exercise therapy in hip abduction/adduction, hip flexion/extension, exercises with low resistance (>12-15 repetitions37), or no resistance and exercises performed in water when sutures had been removed. Each session lasted 1 hour and was performed 5 days a week for 4 weeks.

SUMMARY:
The aim of the study is to improve hospital treatment and rehabilitation of patients with hip arthroplasty to help the patients to regain functional ability in the shortest possible time, and reduce hospital and rehabilitation time to save costs for the patient and society.

Optimal reconstruction of the hip joint and the effect of an intensive physical training programme are compared to conventional rehabilitation programmes.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis
* Unilateral osteoarthritis
* Age below 65 yrs
* ASA group 1-2

Exclusion Criteria:

* Pregnancy
* Age below 18 yrs
* Cardiovascular disease
* Diseases in the musculoskeletal system that could influence on training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hoff, prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Faculty of Medicine, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Husby VS, Helgerud J, Bjorgen S, Husby OS, Benum P, Hoff J. Early maximal strength training is an efficient treatment for patients operated with total hip arthroplasty. Arch Phys Med Rehabil. 2009 Oct;90(10):1658-67. doi: 10.1016/j.apmr.2009.04.018. PMID 19801053